CLINICAL TRIAL: NCT00492635
Title: A Randomized, Double-blind, Double-dummy, Multicenter Parallel Group Study to Compare the Tolerability and Efficacy of Once Daily Vardenafil Versus Vardenafil PRN Versus Placebo in Men Immediately After Nerve-sparing Prostatectomy for Improving Erectile Function
Brief Title: Study to Compare the Tolerability and Efficacy of Once Daily Vardenafil vs Vardenafil PRN vs Placebo in Men Immediately After Nerve-sparing Prostatectomy for Improving ED
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 11336; 2004-002172-42 (EudraCT Number)
Record Dates: First submitted 2007-06-26; First posted 2007-06-27 (Estimated); Last update posted 2014-10-28 (Estimated); Status verified 2014-10

CONDITIONS: Erectile Dysfunction; Sexual Dysfunction, Physiological
MeSH Terms: conditions — Erectile Dysfunction; Sexual Dysfunction, Physiological | interventions — Vardenafil Dihydrochloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (3):
- Arm 1 (Experimental)
  Interventions: Drug: Levitra (Vardenafil, BAY38-9456)
- Arm 2 (Experimental)
  Interventions: Drug: Levitra (Vardenafil, BAY38-9456)
- Arm 3 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Levitra (Vardenafil, BAY38-9456) — 9 months DAILY dosage (double blind) 2 months single-blind placebo wash-out period (subject only is blinded) 2 months open-label PRN treatment with active medication
  Arms: Arm 1
Drug: Levitra (Vardenafil, BAY38-9456) — 9 months PRN dosage (double blind) 2 months single-blind placebo wash-out period (subject only is blinded) 2 months open-label PRN treatment with active medication
  Arms: Arm 2
Drug: Placebo — 9 months placebo (double blind)2 months single-blind placebo wash-out period (subject only is blinded)2 months open-label PRN treatment with active medication
  Arms: Arm 3

SUMMARY:
A study to assess the efficacy of vardenafil, taken as a tablet both nightly or 'as needed' (immediately before intended sexual activity) compared to placebo, to evaluate its tolerability and if it can help in recovery of erections after a nerve sparing radical prostatectomy.

ELIGIBILITY:
Inclusion Criteria:

At Screening

* Males 18-64 years of age
* Scheduled to undergo bilateral nerve-sparing radical retropubic BNSRRP, as selected according to the investigator's usual clinical practice
* Surgery scheduled within about 1 month of screening (Visit 1)
* Expressed an interest in resuming sexual activity as soon as possible after prostatectomy
* Heterosexual relationship
* No pre-operative erectile dysfunction:
* International Index of Erectile Function (IIEF) Erectile Function Domain Score score EF domain =26 at screening without any therapy/devices for improvement of erections
* No perforation of the prostate capsule by tumor

At Randomization:

Before being randomized subjects must still be meeting all Screening Inclusion Criteria, as well as the following criteria:

* bilateral nerve-sparing during the retropubic prostatectomy documented on the operating report
* BNSRRP occurred within approximately 1 month post screening (Visit 1)
* No perforation of the prostate capsule by tumor:

No positive tumor margins confirmed after surgery: =T2 stage on pathology report from the surgery

Exclusion Criteria:

* Subjects who are taking nitrates or nitric oxide donors
* Subjects who are taking the following inhibitors of cytochrome P 450 CYP 3A4: very potent HIV protease inhibitors (ritonavir, indinavir), the anti-mycotic agents itraconazole and ketoconazole (topical forms are allowed) or erythromycin
* Known hypersensitivity to Vardenafil
* Presence of significant penile anatomical abnormalities (e.g. penile fibrosis or Peyronie's disease)
* History of retinitis pigmentosa
* Unstable angina pectoris
* History of myocardial infarction, stroke or life-threatening arrhythmia within the prior 6 months
* Severe chronic or acute liver disease
* Symptomatic postural hypotension in the past 6 months
* NYHA Class III or IV heart failure
* Life expectancy <3 years
* Clinical diagnosis of significant untreated sleep apnea or working night shifts (e.g. 23:00h to 7:00 h)
* Anti-androgens use
* Residual prostate cancer, or requirement for radiotherapy or ADT after surgery

Ages: 18 Years to 64 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 628 (Actual)
Dates: Start 2004-12; Primary Completion 2007-09 (Actual); Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
Determine whether early, NIGHTLY dosing with vardenafil Significantly improves recovery of erectile function after surgery as compared to placebo, and whether early PRN dosing with vardenafil also improves recovery of function as compared to placebo | 9 months

SECONDARY OUTCOMES:
Assess whether early dosing of either NIGHTLY or PRN vardenafil over 9 months, followed by 2 months of withdrawal, increases efficacy of subsequent PRN use significantly better than placebo | 13 months

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (78):
- United States (11):
  - Laguna Hills, California
  - Jeffersonville, Indiana
  - Des Moines, Iowa
  - Jackson, Mississippi
  - Poughkeepsie, New York
  - Cincinnati, Ohio
  - Columbus, Ohio
  - Oklahoma City, Oklahoma
  - Lancaster, Pennsylvania
  - Providence, Rhode Island
  - Spokane, Washington
- Austria (2):
  - Salzburg, Salzburg
  - Graz, Styria
- Belgium (5):
  - Bruxelles - Brussel
  - Edegem
  - Hasselt
  - Leuven
  - Liège
- Canada (10):
  - Calgary, Alberta
  - Edmonton, Alberta
  - Barrie, Ontario
  - London, Ontario
  - Oakville, Ontario
  - Toronto, Ontario
  - Chicoutimi, Quebec
  - Fleurimont, Quebec
  - St. John's
  - Victoria
- Finland (2):
  - Oulu
  - Tampere
- France (5):
  - Carpentras
  - Lille
  - Lyon
  - Nîmes
  - Saint-Genis-Laval
- Germany (11):
  - Mannheim, Baden-Wurttemberg
  - Tübingen, Baden-Wurttemberg
  - München, Bavaria
  - Weiden, Bavaria
  - Hamburg, Hamburg
  - Offenbach, Hesse
  - Braunschweig, Lower Saxony
  - Osnabrück, Lower Saxony
  - Dortmund, North Rhine-Westphalia
  - Herne, North Rhine-Westphalia
  - Leverkusen, North Rhine-Westphalia
- Italy (6):
  - Bari
  - Florence
  - Genova
  - Milan
  - Napoli
  - Trieste
- Netherlands (3):
  - Leiden
  - Nijmegen
  - Rotterdam
- Norway (2):
  - Moelv
  - Tønsberg
- South Africa (4):
  - Johannesburg, Gauteng
  - Pretoria, Gauteng
  - Pietermaritzburg, KwaZulu-Natal
  - Cape Town, Western Cape
- Spain (5):
  - Barcelona, Barcelona
  - Madrid, Madrid
  - Málaga, Málaga
  - Vigo, Pontevedra
  - Valencia, Valencia
- Sweden (5):
  - Gothenburg
  - Halmstad
  - Lund
  - Skövde
  - Västerås
- Bern, Canton of Bern, Switzerland
- United Kingdom (6):
  - Bath, Avon
  - Bristol, Avon
  - Slough, Berkshire
  - London, London
  - Manchester, Manchester
  - Taunton, Somerset

REFERENCES:
- See also: Click here and search for information of Bayer products for Europe — http://www.clinicaltrialsregister.eu